CLINICAL TRIAL: NCT07282145
Title: A Randomized, Double-blinded, Single/Multiple Dosing, Dose Escalation, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of BCD101 in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetics Study of BCD101 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bichedam Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BCD101
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- SAD-1(Treatment group) (Experimental): 6 Participants in the SAD-1(Treatment group) arm received a single oral dose of BCD101-1(2 sachets).
  BCD101-1 is a low-dose liquid formulation containing 2 g of the active ingredient per 10 g sachet.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Low Dose Liquid Formulation
- SAD-2(Treatment group) (Experimental): 6 Participants in the SAD-2(Treatment group) arm received a single oral dose of BCD101-2(2 sachets).
  BCD101-2 is a high-dose liquid formulation containing 4 g of the active ingredient per 10 g sachet.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 High Dose Liquid Formulation
- SAD-3(Treatment group) (Experimental): 6 Participants in the SAD-3(Treatment group) arm received a single oral dose of BCD101-2(3 sachets).
  BCD101-2 is a high-dose liquid formulation containing 4 g of the active ingredient per 10 g sachet.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 High Dose Liquid Formulation
- SAD-4(Treatment group) (Experimental): 6 Participants in the SAD-4(Treatment group) arm received a single oral dose of BCD101-2(4 sachets).
  BCD101-2 is a high-dose liquid formulation containing 4 g of the active ingredient per 10 g sachet.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 High Dose Liquid Formulation
- MAD-1(Treatment group) (Experimental): 6 Participants in the MAD-1(Treatment group) arm received BCD101-1(1 sachet), administered orally twice daily for 7 consecutive days.
  BCD101-1 is a low-dose liquid formulation containing 2 g of the active ingredient per 10 g sachet.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Low Dose Liquid Formulation
- MAD-2(Treatment group) (Experimental): 6 Participants in the MAD-2(Treatment group) arm received BCD101-2(1 sachet), administered orally twice daily for 7 consecutive days.
  BCD101-2 is a high-dose liquid formulation containing 4 g of the active ingredient per 10 g sachet.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 High Dose Liquid Formulation
- MAD-3(Treatment group) (Experimental): 6 Participants in the MAD-3(Treatment group) arm received a combination of BCD101-1(1 sachet) and BCD101-2(1 sachet), administered orally twice daily for 7 consecutive days.
  BCD101-1 is a low-dose liquid formulation containing 2 g of the active ingredient per 10 g sachet, while BCD101-2 is a high-dose liquid formulation containing 4 g of the active ingredient per 10 g sachet.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Low + High Dose Liquid Formulation
- SAD-1(Placebo group) (Experimental): 2 Participants in the SAD-1(Placebo group) arm received a single oral dose of BCD101-P(2 sachets).
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-1, containing no active ingredient.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- SAD-2(Placebo group) (Experimental): 2 Participants in the SAD-2(Placebo group) arm received a single oral dose of BCD101-P(2 sachets).
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-2, containing no active ingredient.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- SAD-3(Placebo group) (Experimental): 2 Participants in the SAD-3(Placebo group) arm received a single oral dose of BCD101-P(3 sachets).
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-2, containing no active ingredient.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- SAD-4(Placebo group) (Experimental): 2 Participants in the SAD-4(Placebo group) arm received a single oral dose of BCD101-P(4 sachets).
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-2, containing no active ingredient.
  This study was conducted as a randomized, double-blinded, placebo-controlled, oral, single-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- MAD-1(Placebo group) (Experimental): 2 Participants in the MAD-1(Placebo group) arm received BCD101-P(1 sachet), administered orally twice daily for 7 consecutive days.
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-1, containing no active ingredient.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- MAD-2(Placebo group) (Experimental): 2 Participants in the MAD-2(Placebo group) arm received BCD101-P(1 sachet), administered orally twice daily for 7 consecutive days.
  BCD101-P is a placebo liquid formulation identical in appearance and volume to BCD101-2, containing no active ingredient.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation
- MAD-3(Placebo group) (Experimental): 2 Participants in the MAD-3(Placebo group) arm received BCD101-P(2 sachets), administered orally twice daily for 7 consecutive days.
  BCD101-P is a placebo liquid formulation identical in appearance and volume to the active formulations, containing no active ingredient.
  The study was conducted as a randomized, double-blinded, placebo-controlled, multiple-dose, dose-escalation trial.
  Interventions: Drug: BCD101 Placebo Liquid Formulation

INTERVENTIONS:
Drug: BCD101 Low Dose Liquid Formulation — [SAD] A liquid formulation of BCD101 containing 2 g of the active ingredient per 10 g sachet, administered orally. Used for single dosing at low concentration.
  [MAD] A liquid formulation of BCD101 containing 2 g of the active ingredient per 10 g sachet, administered orally. Used for multiple dosing at low concentration.
  Arms: MAD-1(Treatment group); SAD-1(Treatment group)
Drug: BCD101 High Dose Liquid Formulation — [SAD] A liquid formulation of BCD101 containing 4 g of the active ingredient per 10 g sachet, administered orally. Used for single dosing at high concentration.
  [MAD] A liquid formulation of BCD101 containing 4 g of the active ingredient per 10 g sachet, administered orally. Used for multiple dosing at high concentration.
  Arms: MAD-2(Treatment group); SAD-2(Treatment group); SAD-3(Treatment group); SAD-4(Treatment group)
Drug: BCD101 Low + High Dose Liquid Formulation — [MAD] A combination of low-dose and high-dose BCD101 liquid formulations, administered orally as separate sachets simultaneously. Used for multiple dosing.
  Arms: MAD-3(Treatment group)
Drug: BCD101 Placebo Liquid Formulation — [SAD Placebo] A placebo liquid formulation matching the appearance and volume of BCD101 sachets, containing no active ingredient. Administered orally. Used for single dosing.
  [MAD Placebo] A placebo liquid formulation matching the appearance and volume of BCD101 sachets, containing no active ingredient. Administered orally. Used for multiple dosing.
  Arms: MAD-1(Placebo group); MAD-2(Placebo group); MAD-3(Placebo group); SAD-1(Placebo group); SAD-2(Placebo group); SAD-3(Placebo group); SAD-4(Placebo group)

SUMMARY:
A randomized, double-blinded, single/multiple dosing, dose escalation Phase 1 clinical trial to evaluate the safety, tolerability, and pharmacokinetic characteristics of BCD101 in healthy adult volunteers.

The primary objectives of this study are to determine:

1. The safety and tolerability of BCD101 in healthy adult volunteers.
2. The pharmacokinetic profile of BCD101 following single and multiple dosing.

A control group is included, and dose cohorts will be compared to assess dose-dependent differences in safety, tolerability, and pharmacokinetics.

Key study activities include:

1. Administration of single and multiple escalating doses of BCD101 and placebo under controlled conditions.
2. Safety and tolerability assessments, including monitoring for serious adverse events and serious adverse drug reactions (Serious AEs/ADRs).
3. Collection of blood samples for pharmacokinetic analysis.

ELIGIBILITY:
1. Inclusion Criteria

   * Healthy adult volunteers aged 19 years or older at screening.
   * Body weight ≥ 50.0 kg and body mass index (BMI) between 18.0 kg/m² and 30.0 kg/m² at screening.

     * BMI (kg/m²) = weight (kg) / {height (m)}²
   * No congenital or chronic medical conditions requiring treatment, and no pathological signs or findings upon medical examination.
   * Clinical laboratory tests, vital signs, physical examination, and 12-lead electrocardiogram (ECG) results at screening indicate suitability for participation based on the characteristics of the investigational medicinal product.
   * Fully understood the detailed explanation of this clinical trial, voluntarily agreed to participate, and provided written informed consent agreeing to comply with study requirements during the trial period.
2. Exclusion Criteria

   * History or current clinically significant liver, kidney, neurological, psychiatric, respiratory, endocrine, hematological, neoplastic, genitourinary, cardiovascular, gastrointestinal, or musculoskeletal disorders.
   * Female subjects who are pregnant (urine hCG positive) or breastfeeding.
   * History of hypersensitivity (e.g., anaphylaxis, angioedema) or clinically significant allergic reactions to the active ingredient, excipients of the investigational product, or other medications (e.g., aspirin, penicillin antibiotics, macrolide antibiotics).
   * History of gastrointestinal diseases or surgeries that could affect absorption of the investigational drug (e.g., Crohn's disease, ulcers, acute or chronic pancreatitis), except simple appendectomy or hernia surgery.
   * Clinically significant abnormalities on 12-lead ECG at screening, including:

     * QTc interval > 450 ms (males) or > 470 ms (females)
     * PR interval > 200 ms
     * QRS duration > 120 ms
   * Clinically significant laboratory abnormalities at screening, including:

     * Liver function tests (AST, ALT, ALP, γ-GT, total bilirubin) exceeding twice the upper limit of normal.
     * Serum creatinine outside the reference range or estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m² as calculated by the CKD-EPI formula.
   * History of substance abuse or positive urine drug screening for abuse substances.

Vital signs at screening after at least 3 minutes of rest in a seated position meet any of the following:

* Systolic blood pressure ≤ 90 mmHg or ≥ 150 mmHg
* Diastolic blood pressure ≤ 60 mmHg or ≥ 100 mmHg
* Pulse rate ≤ 40 bpm or ≥ 100 bpm

  * Evidence of orthostatic hypotension at screening.
  * Use of enzyme-inducing or inhibiting drugs such as barbiturates within 1 month prior to first dosing.
  * Abnormal diet or consumption of foods that could affect drug absorption, distribution, metabolism, or excretion.
  * Use of prescription or herbal medications that may affect the investigational product's characteristics within 2 weeks prior to first dosing, or over-the-counter drugs or dietary supplements within 10 days prior to first dosing (except when judged by the investigator not to affect the pharmacokinetics of the investigational product).
  * Participation in another clinical trial with investigational drug administration within 6 months prior to first dosing (the end date of participation is calculated as the day after the last dose of the previous trial).
  * Whole blood donation within 2 months prior to first dosing, platelet donation within 1 month prior to first dosing, blood transfusion within 1 month prior to first dosing, or inability to abstain from blood donation from informed consent to PSV.
  * Excessive alcohol consumption (more than 21 units per week; 1 unit = 10 g = 12.5 mL pure alcohol) within 6 months prior to first dosing or inability to abstain from alcohol from informed consent to PSV.
  * Smoking more than 10 cigarettes per day within 3 months prior to first dosing or inability to abstain from smoking from 24 hours prior to first dosing until last blood sampling.
  * Consumption of grapefruit-containing foods within 72 hours prior to first dosing or inability to abstain until PSV.
  * Consumption of caffeine-containing foods or beverages (e.g., coffee, green tea, black tea, carbonated drinks, coffee milk, energy drinks) from 24 hours prior to first dosing until last blood sampling or inability to abstain.
  * Engaging in strenuous exercise exceeding daily activity levels from 48 hours prior to first dosing until PSV or inability to refrain from such exercise.
  * Planning to become pregnant or not using reliable contraception methods (e.g., hormonal contraceptives, intrauterine device, sterilization procedures, barrier methods) for self or partner from informed consent until 90 days after last dose of investigational product.
  * Any other reasons deemed by the investigator to make the subject unsuitable for participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (Single-Ascending Dose, SAD) | Day -1, Day 1, post-study visit (Day 4-7)
  All adverse events occurring during the clinical trial following a single ascending dose of BCD101 will be collected and evaluated for seriousness, severity, and their relationship to the investigational product. Events will be coded using MedDRA System Organ Class and Preferred Term.
  [Unit of Measure] Participants
Physical Examination Abnormalities (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  A complete physical examination will be performed, and findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as abnormalities for this outcome measure. Non-clinically significant deviations (NCS) will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported.
  [Unit of Measure] Participants
Vital signs: Systolic and Diastolic Blood Pressure (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  Systolic and diastolic blood pressure will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] mmHg
Vital signs: Heart Rate (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  Heart rate will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] Beats per minute (bpm)
Vital signs: Body Temperature (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  Body temperature will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] °C
Electrocardiogram (ECG) Abnormalities (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  A standard 12-lead electrocardiogram will be performed, and ECG findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as ECG abnormalities for this outcome measure. Non-clinically significant deviations (NCS) from reference ranges will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported.
  [Unit of Measure] Participants
Laboratory Abnormalities (SAD) | Screening, Day -1, Day 1, post-study visit (Day 4-7)
  Clinical laboratory tests will include hematology, clinical chemistry, urinalysis, serology, and urine drug screening. Laboratory findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as laboratory abnormalities for this outcome measure. Non-clinically significant deviations (NCS) from reference ranges will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported.
  [Unit of Measure] Participants
Number of Participants With Adverse Events (MAD) | Day -1 through Day 7, and post-study visit (Day 8-12)
  All adverse events occurring during the clinical trial following a multiple ascending dose of BCD101 will be collected and evaluated for seriousness, severity, and their relationship to the investigational product. Events will be coded using MedDRA System Organ Class and Preferred Term.
  [Unit of Measure] Participants
Physical Examination Abnormalities (MAD) | Screening, Day -1, Day 1, Day 7, post-study visit (Day 8-12)
  A complete physical examination will be performed, and findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as abnormalities for this outcome measure. Non-clinically significant deviations (NCS) will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported.
  [Unit of Measure] Participants
Vital signs: Systolic and Diastolic Blood Pressure (MAD) | Screening, Day -1 through Day 7, and post-study visit (Day 8-12)
  Systolic and diastolic blood pressure will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] mmHg
Vital signs: Heart Rate (MAD) | Screening, Day -1 through Day 7, and post-study visit (Day 8-12)
  Heart rate will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] Beats per minute (bpm)
Vital signs: Body Temperature (MAD) | Screening, Day -1 through Day 7, and post-study visit (Day 8-12)
  Body temperature will be measured after at least three minutes of rest in the seated position.
  [Unit of Measure] °C
Electrocardiogram (ECG) Abnormalities (MAD) | Screening, Day -1, Day 1, Day 7, post-study visit (Day 8-12)
  A standard 12-lead electrocardiogram will be performed, and ECG findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as ECG abnormalities for this outcome measure. Non-clinically significant deviations (NCS) from reference ranges will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported.
  [Unit of Measure] Participants
Laboratory Abnormalities (MAD) | Screening, Day -1, Day 1, Day 6-7, post-study visit (Day 8-12)
  Clinical laboratory tests will include hematology, clinical chemistry, urinalysis, serology, and urine drug screening. Laboratory findings will be categorized as normal, not clinically significant (NCS), or clinically significant (CS). Only clinically significant (CS) findings will be classified as laboratory abnormalities for this outcome measure. Non-clinically significant deviations (NCS) from reference ranges will not be classified as abnormalities. The number of participants with clinically significant abnormalities will be reported. [Unit of Measure] Participants

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: Maximum Plasma Concentration (Cmax) (SAD) | Day 1 (pre-dose through 12 hours post-dose)
  Cmax will be determined using non-compartmental analysis following a single ascending dose of BCD101.
  [Unit of Measure] ng/mL
Pharmacokinetic Parameters: Area Under the Concentration-Time Curve (AUC₀-t) (SAD) | Day 1 (pre-dose through 12 hours post-dose)
  AUC₀-t will be calculated using non-compartmental analysis following a single ascending dose of BCD101.
  [Unit of Measure] ng·h/mL
Pharmacokinetic Parameters: Area Under the Concentration-Time Curve Extrapolated to Infinity (AUCinf) (SAD) | Day 1 (pre-dose through 12 hours post-dose)
  AUCinf will be calculated from the concentration-time curve following a single ascending dose of BCD101.
  [Unit of Measure] ng·h/mL
Pharmacokinetic Parameters: Time to Maximum Plasma Concentration (Tmax) (SAD) | Day 1 (pre-dose through 12 hours post-dose)
  Tmax will be derived from the plasma concentration-time profile following a single ascending dose of BCD101.
  [Unit of Measure] Hour (h)
Pharmacokinetic Parameters: Terminal Elimination Half-Life (t1/2) (SAD) | Day 1 (pre-dose through 12 hours post-dose)
  Terminal elimination half-life will be estimated from the terminal phase of the concentration-time curve following a single ascending dose of BCD101.
  [Unit of Measure] Hour (h)
Pharmacokinetic Parameters: Maximum Plasma Concentration at Steady State (Cmax,ss) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 5 (pre-dose), Day 6 (pre-dose), Day 7 (pre-dose through 12 hours post-dose)
  Cmax,ss will be measured at steady state during multiple ascending dosing (Day 1-7).
  [Unit of Measure] ng/mL
Pharmacokinetic Parameters: Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau,ss) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 5 (pre-dose), Day 6 (pre-dose), Day 7 (pre-dose through 12 hours post-dose)
  AUCtau,ss will be calculated at steady state during multiple ascending dosing (Day 1-7).
  [Unit of Measure] ng·h/mL
Pharmacokinetic Parameters: Area Under the Concentration-Time Curve Extrapolated to Infinity at Steady State (AUCinf,ss) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 5 (pre-dose), Day 6 (pre-dose), Day 7 (pre-dose through 12 hours post-dose)
  AUCinf,ss will be calculated from the plasma concentration-time profile extrapolated to infinity at steady state during multiple ascending dosing (Day 1-7).
  [Unit of Measure] ng·h/mL
Pharmacokinetic Parameters: Time to Maximum Concentration at Steady State (Tmax,ss) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 5 (pre-dose), Day 6 (pre-dose), Day 7 (pre-dose through 12 hours post-dose)
  Tmax,ss will be derived from the plasma concentration-time profile at steady state during multiple ascending dosing (Day 1-7).
  [Unit of Measure] Hour (h)
Pharmacokinetic Parameters: Terminal Elimination Half-Life at Steady State (t1/2,ss) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 5 (pre-dose), Day 6 (pre-dose), Day 7 (pre-dose through 12 hours post-dose)
  The terminal elimination half-life at steady state will be estimated from the terminal phase of the plasma concentration-time curve during multiple ascending dosing (Day 1-7).
  [Unit of Measure] Hour (h)
Pharmacokinetic Parameters: Accumulation Ratio (Rac) (MAD) | Day 1 (pre-dose through 12 hours post-dose), Day 7 (pre-dose through 12 hours post-dose)
  Rac will be calculated as the ratio of steady-state to single-dose exposure during multiple ascending dosing (Day 1-7).

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea